CLINICAL TRIAL: NCT02365623
Title: An Open-Label Study to Explore the Safety, Efficacy and Pharmacokinetics of TMC207 in Japanese Patients With Pulmonary Multi-Drug Resistant Tuberculosis (MDR-TB)
Brief Title: An Exploratory Study of TMC207 in Japanese Participants With Pulmonary Multi-Drug Resistant Tuberculosis (MDR-TB)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Pharmaceutical K.K. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR105158; TMC207TBC2001 (Other: Janssen Pharmaceutical K.K.)
Record Dates: First submitted 2015-02-13; First posted 2015-02-19 (Estimated); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Tuberculosis, Multidrug-Resistant
Keywords: Pulmonary Multi-Drug Resistant Tuberculosis (MDR-TB); TMC207; Bedaquiline
MeSH Terms: conditions — Tuberculosis, Multidrug-Resistant | interventions — bedaquiline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (1):
- TMC207 (bedaquiline) + Background Regimen (BR) (Experimental): Participants will receive TMC207 (bedaquiline) 400 milligram (mg) as 4*100 mg tablets once daily 2 weeks (14 days). From Week 3, participants will receive 200 mg (2 tablets) TMC207 (bedaquiline) 3 times a week up to Week 24 along with background regimen (BR). Based on the discussion with the Pharmaceuticals and Medical Devices Agency (PMDA), the extension of 24-week TMC207 treatment with BR drugs may occur up to Week 48, under certain circumstances, such that many BR drugs which are susceptible at the beginning of the Treatment Phase show resistance during the Treatment Phase. After TMC207 is stopped, the BR will be continued up to 78 weeks after conversion or 102 weeks after day 1 (what happens first).
  Interventions: Drug: TMC207 (bedaquiline); Drug: Background Regimen (BR)

INTERVENTIONS:
Drug: TMC207 (bedaquiline) — TMC207 (bedaquiline): Participants will receive TMC207 (bedaquiline) 400 milligram (mg) as 4*100 mg tablets once daily 2 weeks (14 days) followed by 200 mg (2 tablets) 3 times a week up to Week 24 along with background regimen (BR). Based on the discussion with the Pharmaceuticals and Medical Devices Agency (PMDA), the extension of 24-week TMC207 treatment with BR drugs may occur up to Week 48, under certain circumstances, such that many BR drugs which are susceptible at the beginning of the Treatment Phase show resistance during the Treatment Phase.
  Other Names: Bedaquiline
Drug: Background Regimen (BR) — Participants will receive anti-bacterial tuberculosis drugs (pyrazinamide [PZA], ethambutol [EB, EMB], streptomycin [SM], kanamycin [KM, KAN], enviomycin [EVM], ethionamide [TH], cycloserine [CS], para-aminosalicylic acid [PAS], amikacin [AMK], levofloxacin [LVFX] and other fluoroquinolone. Other drugs are used less commonly, such as amoxicillin-clavulanate, linezolid and clofazimine based on Investigator's decision twice a week from Day 1 up to 78 weeks after conversion or 102 weeks after day 1 (what happens first).

SUMMARY:
The purpose of this study is to explore safety and efficacy of TMC207 administered as part of a multi-drug regimen for 24 to 48-week treatment in Japanese participants with pulmonary multi-drug resistant tuberculosis (MDR-TB), and to evaluate pharmacokinetics (PK) of TMC207 and its primary metabolite M2.

DETAILED DESCRIPTION:
This is an open-label (everyone know the study intervention), single-arm, multicenter trial to explore safety, efficacy and PK of TMC207 in Japanese participants with pulmonary MDR-TB. The participants will receive TMC207 for 24 weeks in combination with individualized BR drugs selected by the Investigator on Day -1. Participants will primarily be assessed for sputum culture conversion at Week 24. Safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Must have confirmed pulmonary multi-drug resistant tuberculosis (MDR-TB) infection, which is defined as infection by a strain of M. tuberculosis resistant to both rifampicin and isoniazid (RFP and INH) by previous screening from a TB treatment
* Must have confirmed positive results for acid-fast bacilli (AFB) on direct smear examination of expectorated sputum specimen (more than [>] 1+ smear-positive) during the Screening Phase or sputum culture positive for M. tuberculosis within the preceding 3 months
* A women must not be of childbearing potential: postmenopausal or permanently sterilized or otherwise be incapable of pregnancy, or if childbearing potential and practicing a highly effective method of birth control consistent with local regulations regarding the use of birth control methods and a man who is sexually active with a woman of childbearing potential and has not had a vasectomy must agree to use a barrier method of birth control
* Must be willing and able to adhere to the prohibitions and restrictions specified in this protocol
* Must sign an informed consent form (ICF) indicating that he or she understands the purpose of and procedures required for the study and are willing to participate in the study

Exclusion Criteria:

* Has any concomitant severe illness or rapidly deteriorating health condition, including immune deficiency that would make implementation of the protocol or interpretation of the study results difficult or otherwise make the subject a poor candidate for a clinical study
* Has complicated or severe extra-pulmonary manifestations of TB, including central nervous system infection
* Participants with significant cardiac arrhythmia requiring medication
* Participants with the abnormal electrocardiogram (ECG) parameters as defined in protocol
* Has human immuno deficiency virus (HIV) antibody positive during the Screening Phase

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2015-02-18 (Actual); Primary Completion 2018-11-08 (Actual); Study Completion 2018-11-08 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With Sputum Culture Conversion | Week 24
  Sputum culture conversion is defined as 2 consecutive negative cultures from sputa collected at least 25 days apart.

SECONDARY OUTCOMES:
Number of Participants With Multidrug resistant (MDRTB) Outcome | Week 102
  Outcome is defined as, Cured: Participants who completed the study and has been consistently culture-negative (at least 5 consecutive negative cultures) for at least 48 weeks. If only 1 positive culture is reported in that time, participant may still be considered cured, provided that this positive culture is followed by a minimum of 3 consecutive negative cultures. Treatment failure: Participants who completed the study and was not cured. Death: Participants who died during study. Participants reported as dead during survival follow-up before or within Week 126 window were included in this category. Participants reported as dead during after Week 126 window are not included in this category as event occurred after planned duration (126 weeks) of study. Transfer out/Default: Participants who discontinued from study for any reason. Treatment completed: Participants who completed the study but did not meet definition for cure or treatment failure due to lack of bacteriologic results.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutical K.K. Clinical Trial, Study Director — Janssen Pharmaceutical K.K.
Locations (2):
- Japan (2):
  - Kiyose
  - Sakai